CLINICAL TRIAL: NCT03811392
Title: Ultrasound Guided Caudal Block Versus Quadratus Lumborum Block for Inguinal Hernioraphy in Preschool Children.
Brief Title: Ultrasound Guided Caudal Block Versus Quadratus Lumborum Block in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia/Head of Ambulatory surgery and pain clinic., University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050108018(18/12/2018)
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hernioraphy/Caudal block (Active Comparator): patients will receive a caudal block after induction of general anaesthesia.
  Interventions: Procedure: Hernioraphy/Caudal block
- Hernioraphy/Quadratus Lumborum block (Active Comparator): patients will receive ultrasound guided quadrates lumborum block (QL )
  Interventions: Procedure: Hernioraphy/Quadratus Lumborum block

INTERVENTIONS:
Procedure: Hernioraphy/Caudal block — 30 patients will receive a caudal block after induction of general anaesthesia
  Arms: Hernioraphy/Caudal block
Procedure: Hernioraphy/Quadratus Lumborum block — 30 patients will receive ultrasound guided quadrates lumborum block
  Arms: Hernioraphy/Quadratus Lumborum block

SUMMARY:
To compare between caudal block and ultrasound guided Quadratus Lamborum block in reducing postoperative pain, opioid consumption, and recovery time following elective inguinal herniorraphy.

The primary outcome:

• to compare between caudal block and ultrasound guided quadratus lamborum block.

The secondary outcome:

* duration of postoperative analgesia.
* incidence of postoperative complications.

DETAILED DESCRIPTION:
After approval of Ethics Committee of the Faculty of Medicine, and taking a written informed consent from the guardians of each patient, the present study will be carried out in Alexandria Main University Hospitals on 60 patients , aged 2 to 5 years and American Society of Anaesthesiologists (ASA) physical status I or II who will be scheduled for elective inguinal herniorraphy in a randomized double blinded study.

The sample size was calculated by High Institute of Public Health.

Exclusion Criteria:

Infection at the site of needle insertion Neuromuscular disease/damage Anticoagulation or bleeding disorder. Sepsis Allergy to local anaesthetics. Guardians refusal

The patients will be randomly divided by closed envelope technique into two groups:

Group I: 30 patients will receive a caudal block after induction of general anaesthesia.

Group II::Will receive ultrasound guided quadrates lumborum block (QL ) ( posterior transmuscular approach ) using 0.5 mL/kg 0.25% bupivacaine to be applied between the QL muscles and the thoracolumbar fascia. .

METHOD

Preoperative Assessment:

1. History taking
2. Clinical examination
3. Routine laboratory investigations including complete blood picture, bleeding and clotting time, prothrombin time, partial thromboplastin time, blood urea, serum creatinine and fasting blood sugar will be done to every patient.

Pre anaesthetic preparation and premedication

* Nothing per mouth for 6 hours before surgery.
* A peripheral cannula (22 G) will be inserted in all patients.
* Administration 0f 10ml/kg. lactated Ringer's solution.
* All patients will be premedicated with atropine 0,1mg/kg. administered IM to all the patients 30 min prior to surgery.

A multi-channel monitor will be attached to the patient to display:

1. Continuous lead II electro cardiogram (ECG) monitoring.
2. Non-invasive blood pressure measurement (NIBP) mmHg.
3. Arterial oxygen saturation by pulse oximeter (SpO2%).
4. End-tidal capnogram (ETco2).

Induction of anesthesia General anesthesia will be induced with sevoflurane and 50% air in oxygen then IV access will be inserted . Fentanyl will be administered at 1 μg/kg, and a laryngeal mask airway will be used to secure the upper airway. Anaesthesia will be maintained with sevoflurane 2% and 50% air in oxygen.

* All procedures (Caudal , QL) will be performed by the same anaesthetist after placement of the LMA before surgery.
* The patients of both groups were admitted to the ward and receive standard postoperative analgesic regimen composed of regular paracetamol 15mg./kg. every 8hours.

According to the studied group, patients will receive after induction either Group I: caudal block. Group II: Quadratus lamborum block.

Technique:

-For the caudal block, the patients were first inducted by GA and then they were placed in the altered left lateral position. The block site, which was mainly at the sacral hiatus, was sterilized with betadine, and the sacral hiatus between the sacral conui was palpated. Then a 23-gage short needle injection was used with the bevel towards the abdomen to puncture the sacral surface at a 45-degree angle. When the sacrococcygeal ligament seemed to have punctured, the needle was tilted more towards the skin surface and the needle was inserted 2-3 mm deeper. The needle was aspired to check for blood and cerebral spinal fluid extravasations. The loss of resistance was confirmed with air-infusion. Then 0.25% bupivacaine 1 ml/kg was infused. (8,9).

In the QL block group, the probe will be placed anterior and superior to the iliac crest, and the 3 abdominal wall muscles will be visualized. The external abdominal oblique muscle will be followed posterolaterally until the posterior border of the muscle will be identified. When the probe is tilted to the attachment site of both the internal abdominal oblique muscle and the external abdominal oblique muscle over the QL, the midline of the thoracolumbar fascia will be seen as a bright hyperechogenic line. A 22-gauge 80-mm Quincke-type SonoPlex needle (Pajunk, Geisingen,Germany) will be inserted using an in-plane technique. The needle will be directed from anterolateral to posteromedial after making a negative aspiration test with 0.5 mL normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 0.5 mL/kg 0.25% bupivacaine will be applied between the QL muscles and the thoracolumbar fascia(10).

The operation will be planned to begin 7 to 10 minutes after the block is applied , and all patients will be operated on with a standardized technique.

Pain levels will be assessed using a FLACC(11) (Face, Legs, Activity, Cry, Consolability ) behavioral pain assessment scale postoperatively . When the FLACC score is 4 or greater ibuprofen 7mg/kg will be administered orally .

Any complications occurring during the procedure will be recorded and treated :

* Hypotension : In childhood, hypotension can be considered significant when there is 20-30% reduction from baseline in systolic blood pressure ( SBP ) (12) . Treated by administering fluid bolus(13) .
* Bradycardia : Defined as(14):

< 60 bpm in kids 3-7 years old . Treated by 0.01-0.02 mg/kg atropine .

• Nausea and vomiting treated with ondansetron 0.1mg/kg intravenously(15) .

MEASURMENTS:

The following parameters will be measured for all patients:

* Pain levels will be assessed using a FLACC (Face, Legs ,Activity, Cry, Consolability) behavioral pain assessment scale postoperatively after recovery at 30minutes and at 1, 2, 4, 6, 12, and24 hours by the nurses and a second anesthetist will be blinded to groupassignment in the recovery room and the surgical ward .
* Duration of analgesia measured by time from start of the block to the first request for analgesia .
* Total analgesic dose .
* Postoperative complications, such as hypotension, arrhythmia, bradycardia,, nausea, or vomiting .
* Parent satisfaction. Satisfaction levels of the parents will be given verbally as a level from 1 to 10, with the lowest level of satisfaction at a value of 1 and the highest level at 10(16).

A-Haemodynamics

1. Heart rate (beats/minute) and rhythm.
2. Non-invasive mean arterial blood pressure (MABP) in mm Hg. Timing

   * Baseline: before the block.
   * Just after the block.
   * Every 5 min during surgery.
   * Every 2 hour after surgery.

B-Need for intraoperative rescue analgesia:

Adequate intraoperative analgesia was defined by hemodynamic stability, as indicated by the absence of an increase in heart rate or systolic arterial pressure 15% compared with baseline values obtained just before surgical incision. An intraoperative increase in blood pressure (BP) or heart rate (HR) by 15% was defined as insufficient analgesia and was treated with a rescue opioid (fentanyl; 1mcg/kg).

C-Assessment of Postoperative analgesia For postoperative pain evaluation, the pain scores were measured and the facial pain scores were taken 10 min, 30 min and 60 min upon arriving into the PACU. The patients were moved to their wards after 90 min passed in the PACU. At 120 min. post-surgery, the last pain scores were taken. The pain scores were taken when the patient was not crying. If the pain score was over 0.6, then paracetamol 15 mg/kg was infused.

D-Analgesic requirements

* Total dose of analgesics postoperative will be recorded
* Time of first analgesic dose given. E-Incidence of postoperative complications: e.g.: nausea , vomiting and respiratory depression.

ELIGIBILITY:
Inclusion Criteria: Patients , aged 2 to 5 years and American Society of Anaesthesiologists (ASA) physical status I or II who will be scheduled for elective inguinal herniorraphy in a randomized double blinded study.

-

Exclusion Criteria:

Infection at the site of needle insertion Neuromuscular disease/damage Anticoagulation or bleeding disorder. Sepsis Allergy to local anaesthetics. Guardians refusal

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pain. | 24 hours
  FLACC Scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meier DE, OlaOlorun DA, Omodele RA, Nkor SK, Tarpley JL. Incidence of umbilical hernia in African children: redefinition of "normal" and reevaluation of indications for repair. World J Surg. 2001 May;25(5):645-8. doi: 10.1007/s002680020072. PMID 11369993
- [Background] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Background] Johr M. Practical pediatric regional anesthesia. Curr Opin Anaesthesiol. 2013 Jun;26(3):327-32. doi: 10.1097/ACO.0b013e3283606a1e. PMID 23614955
- [Background] Hadzic A, Karaca PE, Hobeika P, Unis G, Dermksian J, Yufa M, Claudio R, Vloka JD, Santos AC, Thys DM. Peripheral nerve blocks result in superior recovery profile compared with general anesthesia in outpatient knee arthroscopy. Anesth Analg. 2005 Apr;100(4):976-981. doi: 10.1213/01.ANE.0000150944.95158.B9. PMID 15781509
- [Background] Ecoffey C. Local anesthetics in pediatric anesthesia: an update. Minerva Anestesiol. 2005 Jun;71(6):357-60. PMID 15886601
- [Background] Willard FH, Vleeming A, Schuenke MD, Danneels L, Schleip R. The thoracolumbar fascia: anatomy, function and clinical considerations. J Anat. 2012 Dec;221(6):507-36. doi: 10.1111/j.1469-7580.2012.01511.x. Epub 2012 May 27. PMID 22630613
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Waldman SD. Caudal epidural nerve block: prone position. In: Atlas of Interventional Pain Management, 2nd edn. Philadelphia: Saunders, 2004 ; 380-92
- [Background] Machotta A, Risse A, Bercker S, Streich R, Pappert D. Comparison between instillation of bupivacaine versus caudal analgesia for postoperative analgesia following inguinal herniotomy in children. Paediatr Anaesth. 2003 Jun;13(5):397-402. doi: 10.1046/j.1460-9592.2003.01080.x. PMID 12791112
- [Background] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Nafiu OO, Voepel-Lewis T, Morris M, Chimbira WT, Malviya S, Reynolds PI, Tremper KK. How do pediatric anesthesiologists define intraoperative hypotension? Paediatr Anaesth. 2009 Nov;19(11):1048-53. doi: 10.1111/j.1460-9592.2009.03140.x. Epub 2009 Oct 1. PMID 19796350
- [Background] Pawar D. Common post-operative complications in children. Indian J Anaesth. 2012 Sep;56(5):496-501. doi: 10.4103/0019-5049.103970. PMID 23293390
- [Background] Chiu SN, Lin LY, Wang JK, Lu CW, Chang CW, Lin MT, Hua YC, Lue HC, Wu MH. Long-term outcomes of pediatric sinus bradycardia. J Pediatr. 2013 Sep;163(3):885-9.e1. doi: 10.1016/j.jpeds.2013.03.054. Epub 2013 Apr 25. PMID 23623512
- [Background] Hohne C. Postoperative nausea and vomiting in pediatric anesthesia. Curr Opin Anaesthesiol. 2014 Jun;27(3):303-8. doi: 10.1097/ACO.0000000000000073. PMID 24722005
- [Background] Liversidge XL, Taylor DM, Liu B, Ling SL, Taylor SE. Variables associated with parent satisfaction with their child's pain management. Emerg Med Australas. 2016 Feb;28(1):39-43. doi: 10.1111/1742-6723.12519. Epub 2015 Dec 20. PMID 26685807